CLINICAL TRIAL: NCT02093182
Title: A Retrospective, Open-Label, Non-Randomized, Study Designed to Evaluate the Correlation of HS-1000 Device Capabilities in the Diagnosis and Assessment of Vasospasm Patients After Sub Arachnoid Hemorrhage
Brief Title: An Innovative Non-invasive Acoustic Approach to Detect and Monitor Cerebral Vasospasm
Status: Withdrawn | Type: Observational
Why Stopped: Agreement not executed between site and sponsor
Sponsor: HeadSense Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-007; 0026-14-TLV (Other: Tel Aviv Sourasky Medical Center)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Sub Arachnoid Hemorrhage; Vasospasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The lack of a precise diagnostic technique for cerebral vasospasm associated with traumatic brain injury (TBI) limits the ability to detect and treat this phenomenon. Surveillance Transcranial Doppler ultrasonography (TCD) is the main medical instrument that is utilized to monitor radiographic vasospasm following TBI, yet has its drawbacks such as inaccuracy, highly operator dependent and more.

HS-1000 device, an investigational vasospasm detection device, has the potential to safely diagnose and assess vasospasm with minimal discomfort to patients, allowing a new modality for vasospasm measurement tool.

We aim to evaluate the correlation between the collected and analyzed data from the HS-1000 device and the clinical findings from the TCD tests post-subarachnoid hemorrhage (SAH) patients.

ELIGIBILITY:
Inclusion Criteria:

* SAH patients with a TCD test
* Male or Female in the age range of 18-85 years
* Expected survival > 14 days

Exclusion Criteria:

* Local infection in the ear.
* Pregnant/lactating women
* Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g., mental condition) Note: As the trial does not affect the patient's management, there is no limitation regarding patient's medications, previous or post study procedures, etc.

Enrolled patients treatment will not change due to their participation in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SAH patients with an expected TCD test
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Accuracy analysis | within the first 30 days
  The main goal of the study is to check the feasibility of the HeadSense's non-invasive head monitor to check vasospasm in patients which over went SAH. In order to validate the accuracy of the HeadSense's device, a statistical comparison will be done between the acoustic values from the Headsense device and the TCD outcome.

SECONDARY OUTCOMES:
Safety analysis | within the first 48 hours
  The HeadSense device is non-invasive and radiation free, therefore no major safety issues are expected.
  During the trial, the patient will be monitored to make sure that no danger or damage is caused by the device. Although there is a small chance of adverse events, potential safety issues include:
  * Perforation of the ear drum, caused by inserting the device to the patient's ears
  * Allergic reaction caused by skin contact with the device (the parts that are attached to the skin are taken from an off the shelf stethoscope, so this is very unlikely to happen)
  * Damage to hearing, caused by the generated sound (the sound is 10Db in strength and is being generated for 10 seconds, so hearing damage is very unlikely to happen

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel